CLINICAL TRIAL: NCT00496782
Title: Surrogate Marker For Tropism-A Multi-Center, Open Label, Pilot Study
Brief Title: Multicenter Pilot Study To Define The Marker As An Alternate For Tropism Assay
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: A4001060
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2010-03-19 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Other)
  Interventions: Drug: maraviroc; Procedure: Trofile Assay and HIV RNA quantification assay

INTERVENTIONS:
Drug: maraviroc — Treatment-experienced subjects on failed therapy, with HIV RNA ≥ 1000 copies/mL, are eligible who will receive a tropism assay at screening (Day -14 to 0). Subjects who are eligible will receive maraviroc added to a failing regimen from Day 1 to 14. On day 15, subjects will discontinue the current treatment regimen and begin a new OBT. Subjects with only R5 HIV will continue receiving maraviroc plus OBT. Subjects with non-R5 virus will discontinue receiving maraviroc but continue to receive the new OBT. Investigator selects OBT based on results of phenotype/genotype testing at baseline. The nominal dose for maraviroc is 300 mg BID. The maraviroc dose should be adjusted based on OBT patient is taking. If OBT includes CYP3A4 inhibitor (with or without inducers) maraviroc dose should be 150 mg BID and if OBT includes CYP3A4 inducer (without inhibitors) maraviroc dose should be 600mg BID. If OBT does not include any CYP3A4 inducers or inhibitors maraviroc dose should be 300 mg BID.
Procedure: Trofile Assay and HIV RNA quantification assay — Trofile Assay and HIV RNA quantification assay

SUMMARY:
The purpose of this pilot study is to determine whether there is a correlation between viral load reduction (at Day 4, 7 or 14) following a short course (14 days) of Maraviroc added to a failing regimen, and the R5 result of the TrofileTM assay at screening.

DETAILED DESCRIPTION:
The study A4001060 has been discontinued on April 22, 2008. A review of the poor rate of enrollment has projected difficulties in completing the study in a timely manner, despite the best efforts by the sponsor and the sites. Given the difficulties encountered in this pilot study and the need to conduct an even larger confirmatory study, the decision to discontinue the study has therefore been made. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age (or minimum adult age as determined by local regulatory authorities or as dictated by local law) at the screening visit.
* Have an HIV RNA ≥ 1000 copies/mL, at screening.
* Subjects receiving another investigational antiretroviral compound through participation in a phase 3 or 4 clinical study are eligible to participate in this trial provided.
* That the 2 investigational agents are required to offer the subject a regimen with 2 or 3 active antiretroviral drugs (i.e. one or fewer approved treatment is available to the subject due to prior resistance or intolerance),
* Neither protocol prohibits the use of the other antiretroviral agent, AND the dosing of the two agents when used together is known AND a letter from the Pfizer clinical pharmacologists for maraviroc identifies the dose of maraviroc to be used with other investigational agents.
* Based on screening genotypic resistance testing results the subject must be able to receive at least 3 active drugs other than maraviroc in the new OBT. This is defined as:
* Having three drugs considered susceptible by genotype interpretation (if etravirine will be used, fewer than 3 etravirine resistance mutations will be taken as etravirine susceptibility); or,
* Having two drugs considered susceptible by genotype interpretation (if etravirine will be used, fewer than 3 etravirine resistance mutations will be taken as etravirine susceptibility) and be willing to include raltegravir in the OBT not having used raltegravir in the past.

Exclusion Criteria:

* Potentially life threatening (Grade 4) laboratory abnormality or medical condition.
* Severe hepatic impairment (Child-Pugh classification B or C).
* End stage renal disease or other disease states requiring dialysis therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Hampton, Virginia
- Pfizer Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001060&StudyName=Multicenter%20Pilot%20Study%20To%20Define%20The%20Marker%20As%20An%20Alternate%20For%20Tropism%20Assay

RESULTS

PARTICIPANT FLOW:
Groups:
- CCR5-Tropic HIV-1: Subjects treated with maraviroc in addition to the antiviral regimen they were receiving at the time of Screening (which was a failing regimen) for 14 days (including Day 14). On Day 15, subjects who had CC chemokine receptor 5 (CCR5) human immunodeficiency virus (HIV) 1 (based on Trofile™ assay) continued receiving maraviroc in combination with a new optimized background therapy (OBT) selected by the investigator until End of Study; Maraviroc was dosed orally twice daily (BID) with the total dose adjusted according to the OBT drugs.
- Non-CCR5-Tropic HIV-1: Subjects treated with maraviroc (dosed orally twice daily (BID)) in addition to the antiviral regimen they were receiving at the time of Screening (which was a failing regimen) for 14 days (including Day 14). On Day 15, subjects with non CCR5 HIV 1 or a non reportable Trofile™ assay at Screening had discontinued maraviroc and had a new OBT selected by the investigator until End of Study.
Period: Overall Study
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Started | 9 | 7
Completed | 8 | 5
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1 | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (4.9) | 41.0 (4.8) | 44.0 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Secondary Outcome: Subjects Achieving HIV-1 RNA <400 Copies/mL
Description: Number of Subjects Achieving HIV-1 RNA <400 Copies/mL at each time point
Time Frame: Days 4, 7, 14, 28, and Weeks 8, 12, 18, and 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Subjects Achieving HIV-1 RNA <50 Copies/mL
Description: Number of Subjects Achieving HIV-1 RNA <50 Copies/mL at each time point
Time Frame: Days 4, 7, 14, 28, and Weeks 8, 12, 18, and 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Subjects With Virologic Failure
Description: For this protocol, virologic failure will be confirmed by a repeat viral load test within 2 weeks of first viral load meeting any of the following criteria: 1. Failing to achieve a reduction in HIV-1 RNA > 0.5 log10 copies/mL from baseline by the second viral load determination (unless the viral load is below level of quantification [LOQ]); 2. Experiencing a > 0.5 log10 increase from nadir in HIV-1 RNA after achieving an HIV-1 RNA reduction from baseline > 0.5 log10 copies/mL; or 3. Experiencing an HIV-1 RNA >1000 copies/mL after having achieved an HIV-1 RNA below LOQ.
Time Frame: Baseline up to Week 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Virologic Failure
Description: as for outcome 3
Time Frame: Baseline up to Week 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Lymphocyte Subset CD4 From Baseline
Description: Calculated average of CD4 at Day 7, 14, 28 and Week 24 minus CD4 at Day 1
Time Frame: Day 1 (Baseline), Day 7, 14, 28 and Weeks 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change From Baseline in Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) With R5 & Non-R5 Tropism Results From the Trofile(tm) Assay
Description: Spearman's correlation coefficient to assess percentage of participants achieving HIV-1 RNA with tropism
Time Frame: Baseline, Day 4, 7, 14
Population: Study was canceled: no efficacy data (primary/secondary) was collected per protocol for limited number of patients left in study; only safety data was summarized.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Lymphocyte Subset CD8 From Day 1
Description: Calculated average of CD8 at Day 7, 14, 28 and Week 24 minus CD8 at Day 1
Time Frame: Day 1(Baseline), Day 7, 14, 28 and Weeks 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Lymphocyte Subsets; CD4 and CD8 From Screening.
Description: Calculated avergae of {CD4 or CD8 at Day 1 - CD4 or CD8 at Screening}
Time Frame: Screening (Day -14 to 0), Day 1.
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Detectable Tropism From Screening
Description: Number of subjects who switch their tropism status from screening to Baseline
Time Frame: Screening (Day -21 to 0), Baseline.
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Detectable Tropism From Baseline
Description: Number of subjects who switch their tropism status from Baseline to Days 7, 14, and Week 24/End of Study(EOS)/Discontinuation
Time Frame: Baseline, Day 15 and Week 24/End of Study/Discontinuation
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Detectable Resistance (Genotype) and Susceptibility (Phenotype) to Drugs in the Regimen From Screening
Description: Change in detectable resistance (genotype) and susceptibility (phenotype) to drugs in the regimen from Screening
Time Frame: Screening (Day -21), Baseline (Day 0), Day 14 (after addition of MVC to a failing regimen), Week 24, and time of Virologic Failure.
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Subjects With Susceptibility to Maraviroc
Description: Phenotypic susceptibility to maraviroc
Time Frame: Screening (Day -21 to 0), Day 14, Week 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Gene Sequence in Gp-160, and the V3 Loop From Screening Visit (Day -21 to 0) to Day 14, Time of Virologic Failure (See Section 6.5.1) and Week 24
Description: Change in gene sequence in gp-160, and the V3 loop from Screening visit (Day -21 to 0) to Day 14, time of virologic failure (See Section 6.5.1) and Week 24
Time Frame: Screening (Day -21 to 0), Day 14, time of virologic failure, and Week 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Correlation of Mutations in gp160 and the V3 Loop and Decreased Susceptibility to Maraviroc
Time Frame: Screening (Day -21 to 0), Day 14, time of virologic failure, Week 24
Population: Study was canceled with only 16 subjects of 60 subjects required to enroll.
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CCR5-Tropic HIV-1 | Non-CCR5-Tropic HIV-1
Serious Adverse Events (participants affected / at risk) | 4/9 | 0/7
Other Adverse Events (participants affected / at risk) | 9/9 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCR5-Tropic HIV-1 (N=9) | Non-CCR5-Tropic HIV-1 (N=7)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCR5-Tropic HIV-1 (N=9) | Non-CCR5-Tropic HIV-1 (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Injection Site Pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 0 | 1
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0
Tinea Pedis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Human Papilloma Virus Test Positive (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study terminated prematurely due to slow enrollment. Premature termination of study was not due to any safety concerns. Efficacy data not summarized due to low sample size; only safety was summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.